CLINICAL TRIAL: NCT05069805
Title: Comparison of Erector Spinae Plane Block and Pectoral Nerve Block for Acute and Chronic Pain in Mastectomies Outcomes: a Randomized Clinical Trial
Brief Title: Comparison of Erector Spinae Plane Block and Pectoral Nerve Block for Acute and Chronic Pain in Mastectomies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, Anesthesiology Residency Preceptor, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PECS vs ESP
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Acute Pain; Chronic Pain; Mastectomy
Keywords: Acute pain; Chronic pain; Mastectomy
MeSH Terms: conditions — Acute Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-blind, superiority study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The researcher responsible for the postoperative period, the surgical team and the patients were not aware of the allocated groups. The researcher responsible for the randomization list communicated the researcher responsible for performing the ESP or PECS II block and conducting the anesthesia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS II block group (Active Comparator): Patients in PECS II group will receive general balanced inhaled anesthesia with sevoflurane and fentanyl
  Interventions: Procedure: PECS II block; Procedure: ESP block
- ESP block group (Active Comparator): Patients in ESP group will receive general balanced inhaled anesthesia with sevoflurane and fentanyl
  Interventions: Procedure: PECS II block; Procedure: ESP block

INTERVENTIONS:
Procedure: PECS II block — Patients will receive standard general anesthesia with sevoflurane and fentanyl associated to PECS II block
Procedure: ESP block — Patients will receive standard general anesthesia with sevoflurane and fentanyl associated to ESP block

SUMMARY:
Ultrasound-guided blockage of the erector plane of the spine (known as ESP BLOCK) is a recently described block and a very useful strategy in the perioperative period as it provides effective analgesia in thoracic surgery. Ultrasound-guided type II pectoral nerve block (internationally known by the acronym Pecs II block) is a very useful strategy in the perioperative period because it provides effective analgesia in breast surgeries and can optimize results. The aim of this study is to assess perioperative pain in mastectomies. This is a prospective, randomized, single-blinded study that will compare the effects of spinal erector plane block versus pectoral nerve block in patients scheduled for mastectomy. The ESP group will receive balanced general anesthesia associated with ESP BLOCK with 0.5% ropivacaine guided by ultrasound. The Pecs II group will receive balanced general anesthesia associated with Pecs II block with 0.5% ropivacaine guided by USG.

DETAILED DESCRIPTION:
The integration of ultrasound with anesthesia allowed for greater safety and risk reduction in regional anesthesia, in addition to the possibility of creating new peripheral blocks that contribute to multimodal analgesia, providing greater comfort for patients in the postoperative period. The spinal erector plane block (ESP Block) and type II pectoral nerve block (PECS II block) emerge as yet another analgesia strategy for breast surgeries, as they are less invasive than thoracic epidural anesthesia and paravertebral block thoracic, reducing the risk of complications. The ESP Block was initially described for analgesia in chest surgery and for the management of chronic chest pain. PECS II block was inspired by the infraclavicular approach, and aims at anesthesia of the lateral and medial pectoral nerves, intercostobrachial, 4th, 5th and 6th intercostal nerves and the long thoracic nerves. Both are technically simple and easily reproducible.

Both are safe techniques, easy to reproduce, have a low risk of complications and allow good control of acute perioperative pain. Therefore, our study has as primary objective to compare the quality of perioperative analgesia offered by ESP Block versus PECS II block by intraoperative opioid consumption in oncologic mastectomy.

A pilot study carried out in our service indicated the superiority of PECS II block over ESP block in relation to intraoperative opioid consumption. The proposal is therefore a prospective, randomized, single-blind, superiority study to compare the hypothesis that PECS II is superior to ESP block in oncological mastectomy performed at Hospital de Base do Distrito Federal, Brasília, DF, Brazil.

The patients were randomized 1:1 by a previously generated random list (https://www.randomizer.org). The allocation sequence was kept inaccessible to all investigators during recruitment and treatment. The researcher responsible for the postoperative period, the surgical team and the patients were not aware of the allocated groups. The researcher responsible for the randomization list communicated the researcher responsible for performing the ESP or PECS II block and conducting the anesthesia.

Upon arrival in the operating room, all patients will receive standard monitoring with cardioscopy, pulse oximetry, non-invasive blood pressure and temperature. After venoclysis of the contralateral upper limb to surgery, all patients will receive 0.05 mg/kg intravenous (IV) midazolam, 1mcg/kg fentanyl for anxiolysis, and IV dexamethasone 4 mg. After anxiolysis, blockade will be performed according to the group to which the patient was previously allocated.

All patients will receive general anesthesia, which will be performed with intravenous induction of fentanyl, lidocaine, propofol and rocuronium at the discretion of the anesthesiologist. Anesthesia will be maintained with sevoflurane (approximately 1 to 1.5 minimal alveolar concentration expired fraction, to maintain a bispectral index between 40 and 60). Increases of more than 20% of baseline systolic blood pressure will be interpreted as pain and increments of 1 mcg/kg of fentanyl will be made with each episode, judiciously endorsed by two examiners. Reductions of more than 20% of the systolic arterial pressure or less than 90 mmHg will be treated with ephedrine 5 to 10 mg. Heart rate reductions below 50 bpm associated with a reduction in systolic blood pressure will be treated with 0.5-1 mg atropine.

After sedoanalgesia has been performed, patients allocated to the ESP BLOCK group will receive antisepsis with 70% alcohol at the block puncture site on the ipsilateral side to be operated. Patient will be placed in a seated position with support from assistants. Applied high frequency linear SonoSite M-Turbo® ultrasound probe, protected with a sterile plastic cover. Probe apposition in the paravertebral region identifying the transverse process of the T5 vertebra, the structures of the trapezius, rhomboid and erector spinal muscles, which are arranged in sonoanatomy in this order from the most superficial to the deepest. Insertion of the UniPlex NanoLine® 22Gx50mm needle in plane, towards the transverse process of the vertebra. Viewed the entire path of the needle during puncture. An injection of 30ml of 0.5% ropivacaine was performed between the transverse process and the erector muscles of the spine, observing the dispersion of the local anesthetic in this plane.

After performing sedoanalgesia, patients allocated to Pecs II group will receive antisepsis with 70% alcohol at the puncture site of the breast block to be operated. Patient in supine position with his arm abducted at 90 degrees. Application of a SonoSite M-Turbo® ultrasound high frequency linear probe, protected with a sterile plastic cover. Apposition of the probe in the region inferior to the clavicle, deltopectoral sulcus, will identify the pectoral muscles with the axillary artery and vein that meet at the level of the first rib. Then, the probe will be displaced distally to the space of the 2nd and 3rd rib, identifying the structures of the pectoralis major, pectoralis minor and serratus muscles, which are arranged in the sonoanatomy in this order from the most superficial to the deepest. Insertion of the UniPlex NanoLine® 22Gx50mm needle in plane. Viewed the entire path of the needle during puncture. An injection of 10ml of 0.5% ropivacaine will be performed between the pectoralis major and minor muscles. Progression of the needle to the interfacial plane of the pectoralis minor and serratus anterior muscles with an injection of 20 ml of 0.5% ropivacaine.

Pre, intra and postoperative information will be recorded in a clinical record and intraoperative values of systolic and mean blood pressure, heart rate, expired sevoflurane fraction, perioperative side effects (nausea and vomiting), consumption of anesthetics, analgesics, vasopressors will be recorded , antiemetics, adverse events. Pain will be assessed by the numerical scale of pain at rest and under exertion (END, ranging from 0 to 10, zero being verified when the patient is without pain and ten, with maximum or unbearable pain) at arrival and discharge of the post-anesthesia care unit, 12 hours and 24 hours after surgery. Rescue medications will be noted in the amount and time of the first dose requested, if any.

During the first 24 hours after surgery, patients who present moderate pain (above 2 by END) will receive as their first analgesic 1g intravenous Dipyrone, every 6 hours. As a second analgesic, in case of persistent pain, tramadol 100mg intravenously, every 6 hours. Patients who experience nausea and/or vomiting will receive 8 mg intravenous ondansetron every 8 hours. The occurrence of adverse events, the length of stay in the PACU and the length of hospital stay will be recorded.

After hospital discharge, in the sixth month after surgery, patients were interviewed using a structured questionnaire. Specifically, an investigator blinded to treatment allocation assessed patient-reported outcomes over the telephone. To determine the prevalence of chronic pain, "yes" or "no" dichotomous questions were used. In case of a positive response, patients were asked to provide detailed information about pain and/or discomfort. Participants then completed the Douler Neuropathique 4 (DN4) questionnaire and the Short Form McGill Pain Questionnaire (SF-MPQ).

Based on data from our previous trial and a pilot study involving 26 participants, we estimated that the proportion of patients consuming fentanyl would be approximately 30% in the PECS-II group. The pilot study indicated an increased risk of fentanyl consumption among patients undergoing ESP, whose magnitude was compatible with a relative risk of 2.0. Thus, considering that the proportion of participants using tramadol would be approximately 60% in the ESP group, a total of 84 participants (42 per group) yielded 80% power to detect this difference between groups at an alpha level of 5% (two tails, two-sample proportions test). The number of participants per group was increased to 92 (46 participants per group) to allow for a 10% dropout rate.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, aged between 18 and 70 years, electively scheduled for mastectomy at Hospital Regional de Sobradinho and Hospital de Base do Distrito Federal;
* American Society of Anesthesiology (ASA) physical status I, II or III

Exclusion Criteria:

* Patient with severe heart disease;
* Patient with severe liver disease;
* Patient with severe kidney disease;
* Patient with a neurological disease;
* Use of psychoactive drugs;
* Pregnant women;
* Patients with allergies to any medication used in the study;
* Patients with chronic pain;
* Patients who refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Analgesic consumption during surgery | During the surgery
  The amount of opioid analgesics consumed during surgery

SECONDARY OUTCOMES:
Anesthetics consumption during surgery | During the surgery
  The amount of inhaled anesthetics consumed during surgery
Tramadol consumption in post-operative | Within the first 24 hours after surgery
  Qualification of pain assessed by the amount of tramadol required postoperatively and the time to request them
Pain Scores on the Numeric Rating Scale | Within the first 24 hours after surgery
  Quantify pain by Numeric Rating Scale (NRS, ranging from 0 to 10 cm, zero being found when the patient is no pain and ten, with maximum or un bearable pain
Number of participants with adverse events as a measure of safety and tolerability | During the surgery
  Intraoperative hemodynamic stability analysis through the incidence of tachycardia, hypertension, bradycardia, hypotension and consumed vasopressors
Number of participants with adverse events as a measure of safety and tolerability | Within the first 24 hours after surgery
  Incidence of adverse effects such as time of awakening, nausea, vomiting, pruritus, urinary retention, drowsiness
Incidence of post-mastectomy chronic pain syndrome | Sixth month after surgery
  Incidence of post-mastectomy chronic pain syndrome using a questionnaire applied to patients in the late postoperative period
Pain Scores on the Numeric Rating Scale | Sixth month after surgery
  Quantify pain by Numeric Rating Scale (NRS, ranging from 0 to 10 cm, zero being found when the patient is no pain and ten, with maximum or un bearable pain

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Alexandre Avis, MD, Study Director — Hospital de Base do Distrito Federal
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Sinha C, Kumar A, Kumar A, Prasad C, Singh PK, Priya D. Pectoral nerve versus erector spinae block for breast surgeries: A randomised controlled trial. Indian J Anaesth. 2019 Aug;63(8):617-622. doi: 10.4103/ija.IJA_163_19. PMID 31462806